CLINICAL TRIAL: NCT02328768
Title: Compassionate Use of an Intravenous Fish Oil Lipid Emulsion (Omegaven®) for the Treatment of Intestinal Failure Associated Liver Disease in Children
Brief Title: Compassionate Use of Omegaven® for the Treatment of Intestinal Failure Associated Liver Disease in Children
Status: Approved for marketing | Type: Expanded Access
Sponsor: University of Nebraska (Other)
Collaborators: Children's Hospital and Medical Center, Omaha, Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0018-15-FB
Record Dates: First submitted 2014-12-19; First posted 2014-12-31 (Estimated); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Total Parenteral Nutrition-Induced Cholestasis
MeSH Terms: interventions — fish oil triglycerides

STUDY DESIGN:
Expanded Access Types: Individual, Treatment

INTERVENTIONS:
Drug: Omegaven
  Other Names: Intravenous fish oil emulsion

SUMMARY:
The overall purpose of this study is to determine if replacing standard soybean oil based fat emulsions with Omegaven®, a fish oil based fat emulsion, can reverse or prevent the progression of parenteral nutrition associated liver disease. It is a compassionate use protocol for patients who already have significant liver disease related to parenteral nutrition.

DETAILED DESCRIPTION:
Parenteral Nutrition (PN) is a potentially life-saving intervention for children with short bowel syndrome and intestinal failure. Many common neonatal surgical diseases including Necrotizing enterocolitis (NEC), intestinal atresias, and gastroschisis can cause intestinal failure. The recovery from these illnesses often involves prolonged periods of parenteral nutrition. Intestinal Failure Associated Liver Disease (IFALD) is the most prevalent complication of long term parenteral nutrition in children, affecting up to 2/3 of children with short bowel syndrome. Parenteral lipids are an important source of calories in children, and provide essential fatty acids. Development of IFALD is a multifactorial process. Phytosterols contained in soybean based lipid emulsions have been shown to predispose animals to IFALD. Previous studies in children have shown that dosing the soybean based parenteral lipid emulsion at doses greater than 1g/kg/day may contribute to the development of IFALD. It is currently our practice to limit the lipid dose in children at risk of development of IFALD to 1g/kg/day. Despite this, some patients will still develop biochemical evidence of cholestasis and IFALD. Previous studies in humans have shown that children with IFALD who were administered the intravenous fish oil lipid emulsion Omegaven® reduced their serum direct bilirubin levels. This may be due to a reduction in the amount of arachidonic acide derived inflammatory mediators. The investigators hypothesize that administering Omegaven® in place of conventional soybean fat emulsions may reverse or prevent the progression of PN associated cholestasis and thus allow the patient to be maintained on adequate PN until he/she is able to ingest adequate nutrition enterally.

ELIGIBILITY:
Inclusion Criteria:

* Parenteral nutrition (PN) dependent (unable to meet nutritional needs solely by enteral nutrition) and expected to require PN for at least another 30 days.
* Parenteral nutrition associated liver disease (PNALD) as defined as a direct bilirubin ≥ 2mg/dL or by histology and/or currently on Omegaven through another protocol.
* Other causes of liver disease have been excluded. A liver biopsy is not necessary for treatment.
* Exhaustion of standard therapies to prevent the progression of the liver disease including surgical treatment, cyclic PN, avoiding overfeeding, reduction/removal of copper and manganese form PN, advancement of enteral feeding, and the use of ursodiol.

Exclusion Criteria:

* Pregnancy
* Other causes of liver disease
* Enrollment in any other clinical trial involving an investigational agent (unless approved by the designated physicians on the multidisciplinary team)
* The parent/guardian or subject is unwilling to provide consent and assent

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Brian A Jones, MD, Principal Investigator — University of Nebraska Medical Center/Children's Hospital & Medical Center
Locations (1):
- Children's Hospital & Medical Center, Omaha, Nebraska, United States

DOCUMENTS (2):
  • Study Protocol (2017-01-03): https://cdn.clinicaltrials.gov/large-docs/68/NCT02328768/Prot_000.pdf
  • Informed Consent Form (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT02328768/ICF_001.pdf